CLINICAL TRIAL: NCT06864468
Title: A School-Based Partnership With Rural Tribal Schools for the Primary Prevention of Obesity Among American Indian Youth (P2)
Brief Title: Primary Prevention of Obesity in American Indian Youth in Rural Tribal Schools
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Arizona University (Other)
Collaborators: University of Arizona (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Regina Eddie, Associate professor, Co-principal investigator, Northern Arizona University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2235532-4; 2U54CA143925-16 (NIH)
Record Dates: First submitted 2025-02-25; First posted 2025-03-07 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Obesity Prevention; School Wellness Policy
Keywords: school-based; obesity prevention; American Indian children and youth; school wellness policy

STUDY DESIGN:
Intervention Model Description: Year 1 (2025-2026):
  * 4th-grade students at School A and School B will receive the intervention.
  * 4th-grade students at School C and School D will serve as the comparison group (no intervention).
  Year 2 (2026-2027):
  * 4th-grade students at School C and School D will receive the intervention.
  * 4th-grade students at School A and School B will not receive the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Health promotion curricula includes
  Interventions: Behavioral: Health promotion curricula
- Control group (No Intervention): No intervention, usual day to day activities

INTERVENTIONS:
Behavioral: Health promotion curricula — 3-day summer camp and 9-month health promotion curriculum that focuses on physical activity and nutrition
  Arms: Intervention group

SUMMARY:
The goal of this study is to learn if a culturally relevant health promotion curricula prevents obesity among 4th graders in rural tribal schools. The main questions it aims to answer are: 1) Does the health promotion curricula intervention increase diet and physical activity behaviors in 4th grade students? Researchers will compare 4th grade classes who will receive intervention at two intervention schools to 4th grades at two comparison schools who will not receive the intervention.

All participants will have their skin carotenoids assessed using Veggie Meter, complete 24-hour diet recall via telephone, height and weight measured, body composition, answer two surveys about perceptions of their school environment practices and diet patterns at school, wear accelerometers for 7 days

DETAILED DESCRIPTION:
High prevalence of obesity is a serious health concern among American Indian (AI) youth, placing them at disproportionate risk for adult obesity and obesity-driven metabolic diseases such as diabetes, cardiovascular disease, and cancer. Among individuals with diabetes, alarmingly, cancer has become the leading cause of death. This underscores the urgent need to address excess weight in AI youth to protect against obesity-related diseases and cancer. To date, a limited number of intervention studies have been developed to prevent obesity in AI youth with few studies that have used schools for implementation of nutrition and physical activity (PA) interventions. Of these studies none reported significant improvements in weight-related outcomes, but showed modest improvements in knowledge, attitude and behaviors among AI youth related to nutrition and PA. Notably these reviews reported on studies from the late 1990s to early and mid 2000s - a time period before the federal government took action through key federal legislation requiring schools and school districts to provide more healthy foods and promote physical activity. The Child Nutrition and WIC Reauthorization Act of 2004 was the first national policy to require all schools and school districts that receive federal funding under the National School Lunch Program (NSLP) to develop and implement school wellness policies (SWPs). In 2010, the Healthy-Hunger Free Kids Act strengthened nutrition standards to help schools offer healthier school meals and limit access to low nutrient food sources outside the school lunch program such through á la carte, classroom parties, fundraisers, and school events.

Schools in rural tribal communities participate in the NSLP and are an opportune setting to implement obesity prevention measures through school policies, practices and supportive environments. To our knowledge, Dr. Eddie's early work in school-based research is the only published work that assessed school nutrition policies and practices in Navajo Nation schools after the updated school meal and 'competitive' food standards were set forth by the Healthy Hunger Free-Kids Act of 2010. A follow-up pilot research project, using a mixed methods approach, examined the broader school environment beyond nutrition including school wellness policies and practices related to student nutrition, physical activity, other wellness activities. Preliminary conclusions include the following: 1) schools need support to further develop and strengthen wellness policies; 2) strategies to reduce unhealthy snacks and beverages in classrooms, fundraising events are needed; 3) strategies to increase physical activity opportunities are needed; and 4) engaging parents, school boards, communities, and tribal government to support in school wellness efforts.

The goal of P2 is to engage and partner with four primary (K-6) schools on Navajo Nation to support, develop and implement obesity prevention programming. The objectives are to implement an established health promotion curricula among 4th graders after completing formative research to strengthen SWPs at each school, to establish a baseline for each school. We will use a train-the-trainer approach to establish structured lessons and practices, as warranted, for physical education instructors and food service personnel, for example. The health promotion curricula for the students will include culturally tailored health education focused on nutrition and physical activity. We will build on our existing collaborative partnerships with these tribal communities and established relationships with the Navajo Nation tribal schools. We will engage key school personnel for the formative work to better understand current school capacities and resources. Our proposed outcomes will include increased knowledge among students about healthy lifestyle and stronger SWPs that increase opportunities to access fruits and vegetables, increase structured physical activity, and steps to sustain these beyond the 3-year grant period. We hypothesize that participation in our health promotion efforts will strengthen school-specific SWPs, including structured physical activity, and that 4th grade youth will increase their knowledge and exhibit improved behaviors for fruits and vegetables consumption and increased physical activity.

ELIGIBILITY:
Inclusion Criteria: students enrolled in the 4th and 3rd grades at one of the participating schools, has parental consent, ability to attend baseline assessment, and the 3-day summer camp -

Exclusion Criteria: any student not in either the 3rd or 4th grades, and youth who have not completed an application with any known allergies or limitations to physical activity will not be included

-

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | From enrollment to the end of the intervention at 9 months
  Determine height and weight measurements for BMI using calibrated Tanita SC-331S Body Composition Analyzer and SECA Stadiometer
24-hour dietary recalls | From enrollment to the end of the intervention at 9 months
  Diet recalls will be conducted within a 2-week period (2 weekdays and 1 weekend day) using the Nutrition Data System for Research. Trained interviewers will administer the 24-hour recalls over the telephone
Veggie Meter | From enrollment to the end of the intervention at 9 months
  The veggie meter uses a low-energy blue light to quantify changes in skin carotenoid levels using resonance spectrosocopy. The pad of the index finger is scanned.
Physical activity wrist acclerometer (ActiGraph) | From enrollment to the end of the intervention at 9 months
  Participants will wear the device for 7 days and nights to capture moderate and vigorous physical activity and sleep.
Health promotion survey | From enrollment to the end of the intervention at 9 months
  Survey measuring healthy lifestyle behaviors

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gachupin FC, Joe JR. American Indian youth: A residential camp program for Wellness. Journal of Health Disparities Research and Practice 2017; 10(4):152-163